CLINICAL TRIAL: NCT03658122
Title: Integrating Behavioral Treatment in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1301710
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Problem;Behaviour;Child; Parent-Child Relations
Keywords: Parent-Child Care; Parent-Child Relationship; Disruptive Behavior; Brief Intervention
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with waitlist control. The waitlist control group will receive the study treatment after a two-month wait.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent-Child Care Treatment (Experimental): Participants receive PC-CARE treatment immediately following the pre-treatment assessment.
  Interventions: Behavioral: Parent-Child Care
- Waitlist Control then Parent-Child Care (Other): Participants wait approximately 2 months with no intervention before completing another pre-treatment assessment (post-waitlist assessment) and receiving PC-CARE treatment.
  Interventions: Behavioral: Parent-Child Care

INTERVENTIONS:
Behavioral: Parent-Child Care — Parent-Child Care (PC-CARE) is a 6-week parenting intervention for children aged 1-10 years and their caregivers. This behavioral intervention involves weekly behavioral assessments, teaching of new skills, in-the-moment practice using the new skills, and discussion of how to incorporate skills at home.

SUMMARY:
This study seeks to assess the usefulness of Parent-Child Care (PC-CARE), a brief behavioral intervention for children with difficult behaviors. It will test whether PC-CARE can help families who talk to their pediatricians about behavior problems by improving parent-child relationships, decreasing disruptive behaviors, and improving parents' knowledge and use of effective parenting strategies. Pediatricians who observe or are told their 2-10-year-old patients have difficult behaviors, such as aggression, disobedience, tantrums, trouble focusing, and/or angry and irritable behaviors, will refer patients to this study.

At a first assessment, parents will complete questionnaires about the child's behaviors, parents and children will participate in a 12-minute play observation, and children will have their heart rate and blood flow measured during a 6-minute play observation. After this assessment, families will be randomly assigned either to begin PC-CARE right away or to wait about two months to begin PC-CARE.

Those who begin right away will attend weekly one-hour appointments for six weeks. During appointments, parents and children report on difficult behaviors from the week, learn new positive communication, regulation, and behavior management skills, are observed during a 4-minute play observation, are coached to use the skills (i.e., have the therapist tell the parent how to use skills while interacting with the child), and discuss how to incorporate these skills at home. Parents and children are also asked to play together for five minutes daily at home. At the end of the six weeks, parents and children will complete the same assessments they did at the beginning.

Those who wait to begin PC-CARE will be asked to complete the same questionnaires and observations again before beginning PC-CARE. They will then receive the same treatment as families who began PC-CARE right away. All families will be called one- and six- months after ending PC-CARE to complete a brief questionnaire about the child's behaviors.

Main study hypotheses include:

1. Parents' positive communication with children will improve with PC-CARE
2. Parents will report less parenting stress after PC-CARE
3. Parents will report fewer child behavior problems after PC-CARE
4. Children will show lower stress reactivity (heart rate and blood flow) after PC-CARE
5. Parents will report similar levels of child behavior problems one- and six-months after completing PC-CARE

DETAILED DESCRIPTION:
The current study proposes offering Parent-Child Care (PC-CARE; Timmer et al., 2018), a brief (6-session) behavioral intervention, to children from 2-10 years of age within the primary care building with the goal of improving parent-child relationships, decreasing child disruptive behaviors, and improving parents' knowledge and use of effective parenting strategies, as well as better integrating behavioral health treatments within the primary care setting. To assess the acceptability of integrating these services within primary care, the investigators will examine the proportion of families who participate in treatment out of the total number referred, and the proportion of families completing treatment. To determine the efficacy of PC-CARE in meeting treatment goals, this study uses a randomized control trial study design with a PC-CARE treatment group and a waitlist control group. To better understand the effects of the intervention and potential mechanisms related to improvements in children's disruptive behaviors, the study uses multiple assessment modalities, including parent-report questionnaires, behavioral observations, and physiological data during parent-child interactions. The investigators will additionally assess maintenance of treatment gains by conducting follow-up assessments at one- and six-months post-treatment.

The following hypotheses will be tested:

Hypothesis 1: Increase acceptability of integrative primary care.

A. The proportion of families who agree to treatment with be at least 75% of those who are referred, and the retention rate for completing PC-CARE will be at least 90%.

B. Caregiver-child dyads that receive PC-CARE when compared to the waitlist control group will report higher levels of satisfaction with their primary care provider and medical office (as measured by the Pediatrics Satisfaction Survey).

Hypothesis 2: Improve pediatricians' ability to detect child mental health service needs.

A: The total number of referrals per month will increase over the two-year grant period; demonstrating pediatricians' enhanced ability to recognize the need for behavioral services.

Hypothesis 3: Improve parenting skills

A. Caregiver-child dyads that receive PC-CARE when compared to the waitlist control group will show significant increases in positive communication skills (as measured by PC-CARE observational coding) from pre to post treatment.

B. Caregivers that receive PC-CARE will report higher levels of parenting competence (as measured by the Brief Parenting Stress Index [PSI4-SF]) compared to the waitlist control group

Hypothesis 4: Improve child behavioral problems and self-regulation

A. PC-CARE trained parents, compared to the waitlist control group, will report significant decreases in levels of child behavior problems (as measured by the Weekly Assessment of Child Behavior [WACB] and Behavior Assessment Schedule for Children, 3rd Edition [BASC-3]) from pre to post treatment.

B. For children with trauma histories, those who complete PC-CARE with their caregivers, compared to the waitlist control group, will show improvements in trauma symptoms from pre- to post-intervention (as measured by the Early Childhood Traumatic Stress Screen [ECTSS] or the Child and Adolescent Trauma Screener [CATS]).

C. After completing PC-CARE with their caregivers, children will show lower levels of autonomic stress reactivity compared to their pre-treatment levels and compared to the waitlist control group (as measured using the Biopac MP150 acquisition unit).

Hypothesis 5: Maintain positive treatment effects

A. Caregivers will report similar levels of child behavior problems (as measured by the WACB) one and six months after treatment as they did at the post-treatment assessment, indicating the treatment gains were maintained.

Before starting recruitment, the investigators will meet with physicians at the pediatrics clinic to discuss the value of integrated primary care, explain the PC-CARE program, and discuss observed behaviors or parent concerns that would warrant referral to the program, and teach them how to make referrals. The investigators will provide the primary care physician (PCP) with information about our research study and intervention and will educate them on appropriate clients. When a PCP feels a child would meet criteria for this study, the PCP will provide the caregiver with the recruitment flier and ask for consent to provide the client's information to the research team.

Caregivers that consent to participate in this research study will complete the pre-treatment assessment with their children and then be placed in either the waitlist control group or in the treatment group. Those placed in the treatment group will actively participate in 6 weekly sessions of PC-CARE treatment and respond to a one-month and six month follow-up phone call to provide support and check up on the child's functioning. Caregivers placed in the waitlist control group will participate in the pre-treatment assessment and after approximately two months will be contacted to complete another pre-treatment assessment and to participate in 6 weekly sessions of PC-CARE treatment and afterward will respond to a one-month and six month follow up phone call to provide support and check up on the child's functioning.

For the pre-treatment assessment, parents will complete various questionnaires related to child behavior, parenting stress, and satisfaction with the pediatrics clinic. Parents and children will participate in a video-recorded 12-minute observational assessment of parent-child dyads as they play together in three semi-structured play situations that are analogs of typical parent-child interactions. Each of the 4-minute scenarios will be coded in the moment by the therapist, and later by a research assistant who is blind to the dyad's treatment group. While the therapist introduces PC-CARE to the caregiver, a trained researcher will work with the child to acquire cardiac physiological signals. Using a combination of age-appropriate explanations, books, and/or puppets, the researcher will explain how the device listens to the child's heart and how it is attached with stickers. Pediatric-grade adhesive electrodes will be applied to the child's torso and connected to an amplifier to record the signals using flexible wires. Physiological signals will be collected using a Biopac MP150 acquisition unit. The ECG100C amplifier will be used to collect electrocardiogram data. Children will then watch a 2-min neutral film clip in order to collect a resting measure of autonomic activity. Following this, they will complete two challenging tasks. First, children will have 3-minutes to work on a difficult puzzle on their own. Second, children will spend 3-minutes working on a difficult tangram puzzle with their caregivers. The difficulty of the materials will be age-adjusted. At the end of the assessment, the therapist will provide information about PC-CARE, identify treatment goals, and indicate whether the family has been assigned to waitlist control group or the treatment group.

During the treatment phase of this study, parents and children will attend weekly one-hour PC-CARE sessions for six weeks. At the beginning of these sessions, parents will complete a brief measure of child behaviors for the week. Then parents, children, and therapist will discuss behaviors from the week and identify behavioral goals for the session. The therapist will then teach new positive communication, self-regulation, and/or behavior management strategies to the parent and child together. The parent-child dyad will then be observed from behind a two-way mirror while they play for four minutes. The therapist will then coach the parent to use the newly learned skills by speaking to the parent via an ear-piece from behind the mirror. The session ends with the therapist reviewing progress with the parent and child and identifying a plan for incorporating new skills into the home environment. Parents and children are also assigned 'Daily CARE' to spend five minutes playing together daily and to use the new skills throughout the day.

A power analysis showed that in order to detect a large-sized effect (i.e., f=0.40, eta-squared = .138) with a power of 80, which is appropriate for a wait-list control design, this study would need a sample size of at least 25 families per group (Cohen, 1988). With an estimated attrition rate of 10%, the investigators plan to recruit 28 dyads for each group, comparison and control (Total N = 56) over the two-year study period. Information will be entered and stored in a Microsoft Access database, designed to score standardized measures and store all information relevant for data analysis. Standardized measures will be double-entered to ensure accuracy of scoring; reliability estimates will be assessed for all information that is "judged" or "coded." Each dyad (parent and child) will be identified by a unique ID composed of the child/participant's assigned subject identification (ID), the time in treatment (should the child receive PC-CARE more than once), and an indicator of which caregiver at any particular time in treatment is the participant in question (e.g., primary participant is mother, secondary participant is father). Data are stored on a secure University of California Davis Children's Hospital server, which is password-protected and backed up daily. Physiological data will be acquired using a University of California Davis issued laptop computer and identified only with the unique ID. Raw data files will be uploaded to a secure University of California Davis Children's Hospital server.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver-child dyads in which the child has been in the custody or care of the caregiver for at least one month.
* Children at least 2 years old and no older than 11 years.
* Caregivers participating in this study must complete all measures assessing the child's functioning pre-intervention and the behavioral observation.
* Caregiver-child dyads participating in this study must agree to be video-taped.
* The caregiver must be able to read at a 4th grade reading level.

Exclusion Criteria:

* Caregiver-child dyads will be excluded from the study if the child has been in the custody or care of the caregiver less than a month.
* Caregiver-child dyads will be excluded from the study if there were any missing pre-treatment assessment measures.
* Caregiver-child dyads will be excluded from the study if the dyad did not consent to be video-taped.
* Caregiver-child dyads will be excluded from the study if the caregiver is unable to receive treatment in English.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in positive communication skills parents use during observations with children. | 7-16 weeks
  Parents' use of positive communication (PRIDE) skills and statements to avoid (Avoid), as coded with the PC-CARE Observational Coding, will be coded during observations with the child at pre-treatment, each weekly session, and post-treatment.
Changes in child behavior problems and improved adaptive functioning on the Behavior Assessment Schedule for Children, 3rd Edition (BASC-3), a parent-reported measure of child behavior. | 7-16 weeks
  BASC-3 composite scales = Externalizing, Internalizing, Behavioral Symptoms, Adaptive Skills. Subscales = Hyperactivity, Aggression, Conduct Problems, Anxiety, Depression, Somatization, Atypicality, Withdrawal, Attention Problems, Adaptability, Social Skills, Leadership, Activities of Daily Living, Functional Communication. Scores are converted to T-scores. T-scores are standardized, with a mean of 50 and standard deviation of 10. For the behavior problem scales, scores above 60 are considered problematic; for the adaptive scales, scores below 40 are considered problematic.
Changes in child behavior problems on the Weekly Assessment of Child Behavior (WACB), a parent-report measure of child behavior. | 6-8 months
  WACB is a 9-item measure of child behavior plus one item regarding parenting stress. Frequency of behaviors (1=never to 7=almost always) and whether behaviors need to change (1=yes, 0=no) are recorded at pre-treatment, each weekly session, post-treatment, one month post-treatment, and six months post-treatment. The parenting stress severity score has a range of 1-7, with higher number indicating more stress. The parenting stress need to change score is either 0 or 1, with 1 indicating the stress level needs to change. The severity of behavior problems is a total score (sum of the 9 behavior problem frequency scales) with a range of 9-63. The behavior problem need to change score is a total score, with a range of 0-9. For both scales, higher scores indicate more problems.
Changes in parenting stress on the Parenting Stress Index-Short Form, 4th Edition (PSI4-SF), a self-report measure of parenting stress. | 7-16 weeks
  PSI4-SF yields four scales: Parent-Child Dysfunctional Relationship, Difficult Child, Parental Distress, and Total Stress. T-scores are computed for each scale. T-scores are standardized scores, with a mean of 50 and standard deviation of 10. Scores above 60 are considered problematic. Parents complete PSI4-SF at pre-treatment and post-treatment.
Change in children's heart rate variability (HRV) via respiratory sinus arrhythmia (RSA) | 7-16 weeks
  Children are connected via sticky electrodes to an ECG100C amplifier to measure electrocardiogram activity (ECG) in response to difficult tasks. RSA, a measure of HRV, is computed from the ECG signal using computer software and the Biopac MP150. RSA is a frequency measure, with a unit of natural log of ms squared (ln ms^2). The RSA indexes variability in heart rate that occurs in a high frequency range, the range of respiration. This variability is attributed to parasympathetic influence on the heart. RSA will be measured at pre-treatment and post-treatment.
Change in children's heart rate variability (HRV) via Root Mean Square of the Successive Difference (RMSSD) | 7-16 weeks
  Children are connected via sticky electrodes to an ECG100C amplifier to measure electrocardiogram activity (ECG) in response to difficult tasks. RMSSD, a measure of HRV, is computed from the ECG signal using computer software and the Biopac MP150. RMSSD looks at changes in the time between heartbeats. The RMSSD indexes variability in heart rate that occurs in a high frequency range, the range of respiration. This variability is attributed to parasympathetic influence on the heart. RMSSD will be measured at pre-treatment and post-treatment.

SECONDARY OUTCOMES:
Proportion of families who agree to treatment | 20 months
  The percentage of families who were referred by pediatricians who agreed to treatment.
Treatment retention | 20 months
  Percentage of families who agree to and begin services who complete the 6th session of PC-CARE.
Reductions in child trauma symptoms by the Early Childhood Traumatic Stress Screen (ECTSS), a parent-report measure of children's trauma exposure and trauma-related symptoms. | 7-16 weeks.
  Parents of 2-6-year-olds will complete the ECTSS. Parents indicate whether or not children experienced any of 11 traumatic events, then indicate whether or not (1=yes, 0=no) children display 17 symptoms indicative of posttraumatic stress disorder. The ECTSS yields a total number of traumatic events (range = 0-11; higher scores indicate more traumatic experiences) and a total trauma score (range = 0-17, higher scores indicate more trauma symptoms). Measures will be completed at pre-treatment and post-treatment.
Changes in child trauma symptoms by Child and Adolescent Trauma Screen (CATS), a parent-report measure of trauma experiences and trauma-related symptoms | 7-16 weeks.
  Parents of 7-10-year-olds will complete the CATS. Parents indicate whether or not children experienced any of 11 traumatic events, indicate how often (0=never to 3=almost always) children display 20 symptoms indicative of posttraumatic stress disorder, and indicate whether or not (yes=1, no=0) those problems interfere in 5 areas of functioning. The CATS yields a total number of traumatic events (range = 0-11; higher scores indicate more traumatic experiences), a total trauma score (range = 0-60, higher scores indicate more trauma symptoms), and a functional impairment score (range = 0-5, higher scores mean more impairment). Measures will be completed at pre-treatment and post-treatment.
Satisfaction with pediatrics clinic will change by Pediatrics Satisfaction Survey | 7-16 weeks
  Parents answer 8 questions about their satisfaction with their pediatrician and pediatrics clinic (1= strongly disagree to 6 = strongly agree). Measure will be completed at pre-treatment and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brandi N Hawk, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Children's Hospital, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timmer SG, Hawk B, Forte LA, Boys DK, Urquiza AJ. An Open Trial of Parent-Child Care (PC-CARE)-A 6-Week Dyadic Parenting Intervention for Children with Externalizing Behavior Problems. Child Psychiatry Hum Dev. 2019 Feb;50(1):1-12. doi: 10.1007/s10578-018-0814-8. PMID 29855819
- [Background] Cohen, J. (1988). Statistical power analysis for the behavioral sciences, 2nd Ed. Lawrence Erlbaum, Hillsdale, NJ